Title: Feasibility of an Educational Intervention for the Prevention of Breast Cancer by

Modifying Risk Behaviors Through a Web Application

Date: November 9, 2020

ID: NCT04396665

Aim: To evaluate the viability of an educational intervention for the prevention of breast cancer risk and the modification of their risk behaviors through the use of a web application in women living in the Principality of Asturias.

Design: pilot test; two arms. The randomization for intervention or control group are doing based on the where the city where the women home is located.

Participants: women aged 235 to 50 without breast cancer diagnosis.

Variables: personal characteristics (age, status, educational level, civil status), MIC index, dietary characteristics, level of physical activity, knowledge related with breast cancer symptoms and risk factors.

Intervention: The Intervention Group received a 6-month intervention using a web-app related. The web-app includes some sections: Information related with breast cancer risk. Breast self-examination. Written text and videos done by a nurse. Physical exercise. Written text and videos done by a physiotherapist. Dietary information. Written text and videos done by a nutrition expert. The Control Group did not receive any intervention.

Data analysis

Initially, the personal characteristics of the sample and the losses produced in the reference population were described. Subsequently, before and after the educational intervention, the variables related to the healthy behaviors under study were described, as well as the variables that referred to knowledge about breast self-examination, risk factors and signs-symptoms of breast cancer. For this, the indices of the descriptive statistics were used: absolute frequencies, percentages, means and standard deviations. The normality of the quantitative variables was determined using the Kolmogorov Smirnov test.

which suggested the use of parametric tests.